CLINICAL TRIAL: NCT03152461
Title: Evaluation of the Clinical Performance of the Quantra System With the Quantra Surgical Cartridge in Adult Patients Undergoing Major Surgical Procedures
Brief Title: Evaluation of the Clinical Performance of the Quantra System With the Quantra Surgical Cartridge
Status: Completed | Type: Observational
Sponsor: HemoSonics LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: HEMCS-008
Record Dates: First submitted 2017-05-09; First posted 2017-05-15 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Blood Loss, Surgical
Keywords: Viscoelastic testing; Coagulation; Quantra; Hemostasis
MeSH Terms: conditions — Blood Loss, Surgical; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Surgical patients: Patients undergoing elective cardiac or vascular surgery involving bypass, or major spine surgery, or surgical patients presenting with acute bleeding in a post-surgical unit.
  Interventions: Diagnostic Test: Quantra System

INTERVENTIONS:
Diagnostic Test: Quantra System — Diagnostic device to monitor coagulation properties of a whole blood sample at the point-of-care.
  Other Names: Quantra Surgical Cartridge

SUMMARY:
This study will evaluate the performance of the Quantra System comprised of the Quantra Hemostasis Analyzer with the Quantra Surgical Cartridge in patients undergoing major surgical procedures specifically, major cardiac and vascular procedures and major orthopedic surgery (primarily complex spine surgeries).

DETAILED DESCRIPTION:
The Quantra System is a fully integrated and automated in vitro diagnostic device which uses SEER Sonorheometry, an ultrasound-based technology, to characterize the viscoelastic properties of a whole blood sample during coagulation. The Quantra Surgical Cartridge was developed to monitor hemostasis during major surgical procedures in adult patients. The cartridge consists of four independent channels each containing different sets of reagents, which provide four measurements performed in parallel yielding six parameters that depict the functional status of a patient's coagulation system.

This multi-center, prospective, observational study will evaluate the performance of the Quantra System as compared to standard coagulation tests and comparable measures determined using the ROTEM Delta.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥18 years
* Subject is scheduled for either 1) cardiac or vascular surgery utilizing cardiopulmonary bypass (CPB) or 2) orthopedic surgery including major deformity correction spine surgery
* Subject has a cardiac assist device and is hospitalized for any procedure
* Subject underwent cardiac, vascular or orthopedic surgery and presents with acute bleeding or suspected hypercoagulability in a post-surgical unit
* Subject is undergoing emergency cardiac, vascular or orthopedic surgery
* Subject is willing to participate and he/she has signed a consent form

Exclusion Criteria:

* Subject is unable to provide written informed consent
* Subject is younger than 18 years
* Subject is incarcerated at the time of the study
* Subject is pregnant
* Subject is currently enrolled in a study that might confound the result of the proposed study
* Subject is affected by a condition that, in the opinion of the surgical team, may pose additional risks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes subjects 18 years or older undergoing a surgical procedure with high risk of intra- or post-operative bleeding. It is anticipated that approximately two-thirds of the enrolled subjects will be cardiac or vascular surgery patients and one-third will be orthopedic surgery patients.
Sampling Method: Non-Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2018-02-09 (Actual); Study Completion 2018-02-09 (Actual)

PRIMARY OUTCOMES:
Comparison of Quantra Clot Time and Clot Stiffness results to standard coagulation test results | Baseline, during surgery, and up to 24 hours post-surgery
  Coagulation function assessed by Quantra and standard coagulation tests
Comparison of Quantra Clot Time and Clot Stiffness results to comparable ROTEM Delta results | Baseline, during surgery, and up to 24 hours post-surgery
  Coagulation function assessed by Quantra and ROTEM Delta

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Maryland Medical Center, Baltimore, Maryland
  - Duke University School of Medicine, Durham, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No